CLINICAL TRIAL: NCT02009761
Title: Safety, Efficacy, Tolerability, Pharmacokinetics and Pharmacodynamics of Open Label Study With Multiple (and for Non Responders) Escalating Subcutaneous Doses of BI 655064 Once a Week in Patients With Chronic Primary Immune Thrombocytopenic Purpura.
Brief Title: Multiple Rising Does Study (Subcutaneous Doses) of BI 655064 in Male and Female Patients With Chronic Primary Immune Thrombocytopenic Purpura (ITP).
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1293.7
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-08

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — BI 655064

ARMS (1):
- BI 655064 120 mg / 180 mg (Experimental): The patients were administered 120 mg BI 655064 solution for subcutaneous injection q1w (once a week) subcutaneously for 4 weeks.
  Patients who showed an increase in platelet count above or equal to 100 x 10^9/L continued treatment with 120 mg BI 655064 solution for subcutaneous injection q1w for additional 8 weeks, followed by 12 weeks of follow-up.
  Patients whose platelet count stayed below 100 x 10^9/L continued treatment for 2 weeks with 180 mg BI 655064 solution for subcutaneous injection q1w followed by 120 mg BI 655064 solution for subcutaneous injection q1w for additional 6 weeks, followed by 12 weeks of follow-up.
  Interventions: Drug: BI 655064

INTERVENTIONS:
Drug: BI 655064 — subcutaneous injection

SUMMARY:
BI 655064 will be administered subcutaneously once weekly in patients with immune thrombocytopenic purpura (ITP) for up to 12 weeks.

ELIGIBILITY:
Inclusion criteria:

Male and female chronic immune ITP patients

Exclusion criteria:

Any treatment of ITP excluded except for a stable dose of corticosteroids (up to 20 mg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2016-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - New York Hospital, Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, multiple dose with dose escalation for non-responders, multiple injection study in patients with chronic primary immune thrombocytopenic purpura.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | BI 655064 120 mg / 180 mg
Started | 6
Completed | 2
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): Included all patients who were dispensed trial medication and were documented to have taken at least one dose of trial medication.
Arm/Group | BI 655064 120 mg / 180 mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Response in Platelet Count
Description: This outcome measure presents number of patients with a response in platelet count. Response was defined as:
  [A] An increase in platelet count by greater than 20 x 10^9/L from baseline at any time-point between Week 1 and Week 12, and [B] Platelet count above 50 x 10^9/L at any time point between Week 1 and Week 12 with no rescue therapy.
  Baseline was defined as the platelet count at Visit 2 before administration of BI 655064. In case the patient fulfilled only one of the conditions, he/she was considered a non-responder.
Time Frame: Up to 12 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BI 655064 120 mg / 180 mg
Number analyzed (Participants) | 6
Participants
  No | 5
  Yes | 1

2. Secondary Outcome: Number of Subjects With Drug-related Adverse Events
Description: Number of participants with investigator defined drug-related adverse events (AEs) is reported.
Time Frame: From first drug administration until end of the Residual Effect Period (REP), up to 6 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BI 655064 120 mg / 180 mg
Number analyzed (Participants) | 6
Participants | 1

3. Secondary Outcome: Number of Patients Reaching the Cut-off Point for Immune Thrombocytopenic Purpura [ITP]
Description: This outcome measure presents the number of patients reaching the cut-off point for ITP, which was defined as: [A] Platelet count ≥ 100 x 10^9/L at any time point between Week 1 and Week 12.
Time Frame: Up to 12 weeks.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BI 655064 120 mg / 180 mg
Number analyzed (Participants) | 6
Participants
  No | 6
  Yes | 0

ADVERSE EVENTS:
Time Frame: From first drug administration until end of the Residual Effect Period (REP), up to 6 weeks.
Description: Treated Set (TS): Included all patients who received trial medication and were documented to have taken at least one dose of trial medication. The safety analysis was pre-specified to display overall, without differentiating treatments (BI 655064 180mg q1w in Weeks 5 and 6, and BI 655064 120mg q1w during the treatment period). The analysis presents the treatment emergent AEs. The on-treatment period: between drug intake until 6 weeks after the last study medication dose.
Arm/Group | BI 655064 120 mg / 180 mg
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 655064 120 mg / 180 mg (N=6)
Conjunctival haemorrhage (Eye disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Hernia (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Haemorrhage (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Trial enrollment was permanently stopped due to low patient enrollment. At the time of termination of enrollment, only 6 patients were entered (only 2 of them completed treatment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.